CLINICAL TRIAL: NCT06953206
Title: SAPIEN Ultra RESILIA Durability EU Registry - The RESOUND-EU Registry
Brief Title: Prospective, Long-term Evaluation of the SAPIEN 3 Ultra RESILIA Valve
Acronym: RESOUND-EU
Status: Not yet recruiting | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Responsible Party: Sponsor
Other Study IDs: RESOUND-EU Registry
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Transcatheter Aortic Valve Replacement (TAVR); Aortic-Stenosis; Aortic Insufficiency; Degenerative Valve Disease
Keywords: TAVR; SAPIEN 3 Ultra RESILIA Valve; S3UR; TAVI; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency | interventions — Replantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVI Patients: Adult patients with severe aortic stenosis undergoing transfemoral TAVI on their native valve with S3UR valve
  Interventions: Procedure: Transcatheter aortic valve (S3UR) replacement (TAVR)

INTERVENTIONS:
Procedure: Transcatheter aortic valve (S3UR) replacement (TAVR) — Elective transfemoral TAVi procedure with S3UR valve.

SUMMARY:
Evaluation of clinical outcomes and valve performance of the SAPIEN 3 Ultra Resilia (S3UR) valve over 10 years.

DETAILED DESCRIPTION:
Transcatheter aortic valve replacement (TAVI) has become the gold standard treatment for moderate-to-high risk elderly patients with severe symptomatic aortic stenosis. Based on the results of randomized trials including low risk patients, this treatment has been progressively applied to younger (in the sixties and seventies) patients with a low co-morbidity burden. Life expectancy in this group is expected to extend beyond 5 years from intervention in the vast majority of patients, and beyond 10 years in a high proportion. Thus, the issue of valve durability has become one of the most important aspects in the TAVI field in recent years. To date, the rates of bioprosthetic valve failure at 8-10 years after TAVI have been consistently <10%, but some studies have shown some degree of valve structural degeneration in close to one third of the patients at 8-year follow-up. This subclinical valve degeneration before the 10-year follow-up landmark would represent the initial step in the process of bioprosthetic valve failure, and further valve degeneration leading to clinical symptoms is likely to occur in a significant proportion of these cases.

This prospective registry will evaluate the clinical outcomes and the valve performance of the SAPIEN 3 Ultra RESILIA valve over 10 years.

ELIGIBILITY:
Inclusion criteria:

* Adult patients (≥18 years)
* Patients with severe aortic stenosis undergoing transfemoral TAVI on their native valve with S3UR valve
* Patient is willing to attend the follow-up visits up to 10 years at the center

Exclusion criteria:

* Lack of written informed consent
* Emergency procedure
* Pregnancy at time of TAVI

Critieria for long-term observation (1y-10y):

* Technical success at exit from procedure room (VARC-3):

  * Freedom from mortality
  * Successful access, delivery of the device, and retrieval of the delivery system
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the device (excluding permanent pacemaker or PTA and stenting without major bleeding) or to a major vascular or access related, or cardiac structural complication
* Absence of the following severe procedural and in-hospital complications (VARC-3 definitions):

  * All stroke
  * Bleeding type 3-4
  * Myocardial infarction
  * Need for a second valve
  * Valve embolization
  * Coronary obstruction
  * Annular rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patiets with severe aortic stenosis planned to undergo TAVR on their native valve with a SAPIEN 3 Ultra RESILIA Valve.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2037-05-30 (Estimated); Study Completion 2037-09-30 (Estimated)

PRIMARY OUTCOMES:
Early Safety | 1-3 months
  Early safety acc. to VARC-3
Device Success | 1-3 months
  Device Success acc. to VARC-3
Bioprosthetic Valve Failure | 3-5 years
  Bioprosthetic valve failure (defined as valve-related mortality OR aortic valve re-operations/re-intervention OR stage 3 hemodynamic valve deterioration (VARC-3))
Bioprosthetic Valve Failure | 9-10 years
  Bioprosthetic valve failure (defined as valve-related mortality OR aortic valve re-operation/re-intervention OR stage 3 hemodynamic valve deterioration (VARC-3))
Structural Valve Deterioration | 9-10 years
  Structural Valve Deterioration ≥ stage 2 (VARC-3)

SECONDARY OUTCOMES:
Hemodynamic Valve Performance | All follow-ups (1-3 month, 1year, 3-5 year, 6-8 year, 9-10 year)
  * Prosthetic valve regurgitation including paravalvular regurgitation
  * Mean transvalvular gradient
  * Max transvalvular gradient
  * Effective orifice area
Bioprosthetic Valve Failure | All follow-ups (1-3month, 1year, 3-5 year, 6-8year 9-10 year)
  Bioprosthetic Valve Failure acc. to VARC-3
Bioprosthetic Valve Dysfunction | All follow-ups (1-3month, 1year, 3-5 year, 6-8year, 9-10 year)
  BVD acc. to VARC-3
Patient reported outcomes | 1-3month, 1+3year Follow Up compared to BL
  Patient reported outcomes using TASQ questionnaire and EQ-5D questionnaire
Cumulated incidence rate BVD or BVF | Up to 10 years
  Cumulated incidence rate (per 100 patient-years) of bioprosthetic valve dysfunction (stage 2 or 3) OR bioprosthetic valve failure up to 10-year follow-up
Clinical Events | All follow-ups (1-3month, 1year, 3-5 year, 6-8year, 9-10 year)
  Clinical events (mortality, stroke, bleeding type 2-4, cardiac rehospitalization, heart failure rehospitalization)
Hemodynamic valve deterioration stage 2 and 3 (VARC-3) | All follow-ups (1-3 month, 1year, 3-5 year, 6-8 year, 9-10 year)
  HVD stage 2 and 3 according to VARC-3 Criteria (moderate and severe HVD).

OTHER OUTCOMES:
Overall kidney function | All follow-ups (1-3month, 1year, 3-5 year, 6-8year, 9-10 year)
  Kidney function assessed through lab values: eGFR in ml/min/1,73m2; creatinine in mg/dl or micromol/l; albumin-to-creatinin-ratio in mg/g; serum calcium in mg/dl or millimol/l ; serum phosphate in mg/dl or millimol/l ; PTH intact in pmol/l, pg/ml or ng/l; Hb in g/l, g/dl, millimol/l
Overall Lipid Status | All follow-ups (1-3month, 1year, 3-5 year, 6-8year, 9-10 year)
  Lipid status assessed through lab values: total cholesterol in mg/dl, millimol/l or micromol/l; LDL in millimol/l or micromol/l; HDL millimol/l or micromol/l;Triglycerides in mg/dl, millimol/l or micromol/l; latest HbA1c in %; Lp(a) in mg/dl or nmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Rudolph, Prof., Principal Investigator — Heart and Diabetes Center North Rhine-Westphalia University Hospital of the Ruhr University Bochum; Michael Joner, Prof, Principal Investigator — German Heart Center
Locations (1):
- Heart and Diabetes Center North Rhine-Westphalia, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
no individual participant data (IPD) will be shard